CLINICAL TRIAL: NCT04327297
Title: Mineral Status in Infants With Cow's Milk Protein Allergy Before and After Receiving Amino Acid-based Formula (AAF)
Brief Title: Mineral Status Ininfants With Cow's Milk Protein Allergy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, israa hosni, Principle investigator, Assiut University
Other Study IDs: Msoiwcmpabaaraabf
Record Dates: First submitted 2020-03-10; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2019-09

CONDITIONS: Cow Milk Allergy
Keywords: Mineral status
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Amino acid-based formula — Amino acid based formula is formula which is used as dietary supplement instead of dairy products in cow's milk allergic infants

SUMMARY:
This study evaluate the mineral status of infants with cow's milk protein allergy which is affected due to the elimination of milk , and the change in this mineral status after receiving amino acid - based formula for 12 weeks.

DETAILED DESCRIPTION:
Introduction Food allergy is defined as an adverse health effect arising from a specific Immune response that occurs following ingestion of a given food . Cow's milk protein (CMP) is the leading cause of food allergy in infants and young children younger than 3 years .Cow's milk contains at least 25 different proteins , all of which may act as antigens .

Prevelance Cow's milk protein allergy (CMPA) does seem to peak in the first year of life, with a prevalence of approximately 2% to 3% in the Infant population . This prevalence then falls to <1% in children 6 years of age and older . A few exclusively breast-fed infants may also develop clinically significant CMPA via dairy protein transfer into human breast milk .

Clinical presentation Manifestations of CMPA may involve many different organ systems mostly the skin and the gastrointestinal and respiratory tract . Skin: Urticaria, Atopic dermatitis. Gastrointestinal: perioral swelling , vomiting, regurgitation, early Satiety, diarrhea (+/-malabsorption or protein loss enteropathy) , failure to thrive, abdominal colic and persistent constipation . Respiratory: runny nose, wheezing and chronic cough. General manifestation: anaphylaxis leading to death in sensitized patient .

Diagnostic procedures Thorough medical history and physical examination. Skin prick test (SPT) and the determination of specific Ig-E in a blood sample. Allergen elimination and controlled challenge procedure. Cow's Milk-related-Symptom-Score (CoMiSS).

A Cow's Milk-related Symptom-Score (CoMiSS) is a score that considers general manifestations ,dermatological and respiratory symptoms.It was developed to be used as an awareness tool for cow's milk related symptoms. It also can be used to evaluate and quantify the evolution of symptoms during therapeutic interventions.

Mineral elements in milk and their nutritional importance There is a sufficient evidence that minerals, both independently or in proper balance with other minerals, have structural, biochemical and nutritional functions that are very important for overall human health, both mental and physical . Furthermore, they act as catalysts for many biological reactions in the body, including muscle contraction, transmission of nerve impulses and utilization of nutrients from food .Many mineral elements are essential in human nutrition: sodium, potassium, chloride, calcium, manganese, selenium, iodine, cobalt .All essential mineral elements can be found in milk because by definition it contains the nutrients required for growth of the young .

Cow milk protein allergy and mineral status

Adequate nutritional intake in infancy is essential to ensure appropriate physiological and mental development .Exclusion diets, in particular cows' milk exclusion diets, have been associated with poor growth in childhood ; as eliminating dairy products in diets of CMP allergic infants ,as well as, coexisting feeding problems ,can result in removing a substantial source of minerals which are involved in essential body functions .This avoidance should ideally be supported by input from an allergy dietitian to monitor and optimise the nutritional content of the diet and to maintain potential growth .

The following treatment options are available for infants with CMPA

1. Hypoallergenic extensively hydrolyzed formulas (eHF) of cow's milk proteins,theses formulas are of choice in patients with CMPA, however, allergic reactions have been reported in children extremely sensitive to cow's milk .
2. Milk derived from purified soya proteins. However, the use of soya is not recommended as a substitute in infants with CMPA under 6 months of age .
3. Milk derived from partial rice protein hydrolysis formulas; they have scant sensitising capacity and do not produce adverse reactions .
4. Free amino acid -based formulas (AAF). Amino acid-based formulas (AAF) Formula containing free amino acids as the only nitrogen source. An (eHF) is recommended for infants with mild to moderate CMA, whereas initiation with an (AAF) is recommended for more severe or complex allergy or when symptom-resolution with (eHF) fails or when (eHF)s are rejected by the patients due to playability problems . Dietary management of CMA with an AAF has been proven to be well-tolerated, effective, and safe; adequate infant growth on an AAF has widely been reported .

ELIGIBILITY:
Inclusion Criteria:

* Infants 1 to 6 months old.
* Diagnosed as cow's milk protein allergic infants according to Cow's Milk-related-Symptom-Score(CoMiSS)(14).

Exclusion Criteria:

* Age: more than 3 month old infants.
* Previously diagnosed to have any gastrointestinal or systemic disease other than CMPA.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants from 1 month to six months
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
blood sample | 1year
  blood sample will be taken to assess/measure the mineral status(including:sodium,potassium,chloride,phosphorus,calcium,magnesium) of infants aged (1-6 months ) diagnosed as cow's milk protein allergy before receiving amino acid - based formula (at start of the study) and after receiving amino acid based formula (for 12 weeks)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Harvey BM, Eussen SRBM, Harthoorn LF, Burks AW. Mineral Intake and Status of Cow's Milk Allergic Infants Consuming an Amino Acid-based Formula. J Pediatr Gastroenterol Nutr. 2017 Sep;65(3):346-349. doi: 10.1097/MPG.0000000000001655. PMID 28604516
- [Result] Koletzko S, Niggemann B, Arato A, Dias JA, Heuschkel R, Husby S, Mearin ML, Papadopoulou A, Ruemmele FM, Staiano A, Schappi MG, Vandenplas Y; European Society of Pediatric Gastroenterology, Hepatology, and Nutrition. Diagnostic approach and management of cow's-milk protein allergy in infants and children: ESPGHAN GI Committee practical guidelines. J Pediatr Gastroenterol Nutr. 2012 Aug;55(2):221-9. doi: 10.1097/MPG.0b013e31825c9482. PMID 22569527
- [Result] Maslin K, Oliver EM, Scally KS, Atkinson J, Foote K, Venter C, Roberts G, Grimshaw KE. Nutritional adequacy of a cows' milk exclusion diet in infancy. Clin Transl Allergy. 2016 Jun 2;6:20. doi: 10.1186/s13601-016-0109-8. eCollection 2016. PMID 27257475
- [Result] Martorell-Aragones A, Echeverria-Zudaire L, Alonso-Lebrero E, Bone-Calvo J, Martin-Munoz MF, Nevot-Falco S, Piquer-Gibert M, Valdesoiro-Navarrete L; Food allergy committee of SEICAP (Spanish Society of Pediatric Allergy, Asthma and Clinical Immunology). Position document: IgE-mediated cow's milk allergy. Allergol Immunopathol (Madr). 2015 Sep-Oct;43(5):507-26. doi: 10.1016/j.aller.2015.01.003. Epub 2015 Mar 20. PMID 25800671